CLINICAL TRIAL: NCT06643767
Title: Evaluation of the Bexa Breast Examination (BBE) As an Effective Solution to Breast Cancer Early Detection
Brief Title: Evaluation of the Bexa Breast Examination
Acronym: BBE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sure, Inc. (Industry)
Collaborators: Hendrick Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Pro00080990
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Bexa; Breast Cancer Screening; Breast Mass Detection; Breast Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: At least 444 women presenting for screening mammograms will undergo the Bexa Breast Exam (BBE). Each woman will receive digital breast tomosynthesis and a BBE on the same day. All women with a positive finding on either digital breast tomosynthesis (mamo-positive), BBE (bexa-positive), or both modalities will undergo a diagnostic ultrasound examination and/or diagnostic mammography of all positive findings.
Masking Description: Open label study; no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Participants (Experimental): Participants scheduled for screening mammography.
  Interventions: Device: Bexa and focus ultrasound

INTERVENTIONS:
Device: Bexa and focus ultrasound — The Bexa exam uses pressure elastography to produce a map of the breast tissue's elasticity to identify any masses. Focused ultrasound is then used to further classify the mass into a BIRADS category.
  Other Names: Bexa Breast Exam

SUMMARY:
Objective:

The "Bexa Breast Exam," or "BBE," for the purposes of this study is defined as the use of a Bexa device in conjunction with a portable, focused ultrasound examination to identify and further evaluate abnormal breast masses including cancer. Commercially, this combination of Bexa plus focused ultrasound is called "Bexa Breast ExamTM," and abbreviated as, "BBE." This study compares the Bexa Breast Exam (BBE) to the standard of care (digital breast tomosynthesis) in detecting masses and as a breast cancer early detection examination.

The specific objectives are:

1. To measure the sensitivity and specificity of BBE as compared to digital breast tomosynthesis in the general population of women over 30 without a history of breast cancer.
2. To measure the sensitivity and specificity of BBE as compared to digital breast tomosynthesis identifying breast masses including cancer in women with dense breasts.
3. To demonstrate the proportion of women receiving a BBE that require additional imaging studies.

Hypothesis:

The purpose of this study is to demonstrate that the Bexa Breast Examination's sensitivity and specificity in identifying abnormal breast masses is comparable to the current accepted standard of care, mammography with tomosynthesis.

DETAILED DESCRIPTION:
Background and Significance:

Breast cancer is the second leading cause of cancer deaths among women in the United States. It is estimated that 287,850 women were diagnosed with breast cancer in 2022, of which 43,250 will die. The current recommended form of screening for breast cancer is mammography, followed by the Clinical Breast Exam, "CBE". However, CBE is subjective, highly variable depending upon training and experience, and lacks the level of sensitivity needed to consistently detect breast masses including cancer.

Mammography can be painful, irradiates the breast, is available primarily in intimidating hospital and/or medical clinic locations and requires physician interpretation. As well, screening mammography results are typically provided to the woman days to weeks after the examination. In a study of 405,191 mammogram examinations, 20% of breast cancers were missed, and 12-14% of examinations had false positives results. A study published in the February 2016 Annals of Internal Medicine posited that among women receiving annual mammography, the radiation exposure caused 246 cancers per 100,000 women over a 10-year period.

Screening mammography is not adopted by between 30% and 60% of American women over 40, with exaggerated challenges to adoption in the African American and Hispanic communities. Mammography is historically not offered to younger women, because it is inaccurate in their denser breast tissue. Over the past decade, the United States Preventive Services Task Force (USPSTF) has acted to limit the use of mammography in women 40-49 due to the high rate of false positive examinations. This has further expanded the population of women at risk for breast cancer without an effective early detection option. While annual screening remains the ideal screening frequency to achieve early detection, screening mammography recommendations from the USPSTF are driving the transition towards mammograms in women over 50 to every 24 to 36 months, primarily as a tactic to limit radiation exposure. However, this approach renders the women between the ages of 40 and 50 with no options for screening and early detection.

Globally, less than 5% of at-risk age women will ever receive screening mammography, primarily due to the expense of the equipment and of the supporting radiology operations.

Efforts must be made to improve the quality and frequency of early detection for all women at risk, particularly for those women who do not readily adhere to breast screening guidelines or for whom screening mammography is no longer a recommended option. An ideal early detection solution should be pain free, radiation free, provide immediate results, and be easily scalable to vulnerable populations. It must have both a low false negative rate and a low false positive rate, generating an acceptably low number of unnecessary referrals for additional and unneeded imaging studies. In order to make an impact upon the global community at-risk, the equipment and its operation must be low-cost, efficient, accessible and scalable. The best cancer screening test is one that patients readily adopt.

Bexa, Inc. has developed a commercially available High-Resolution Pressure Elastography device, the "Bexa™" device, for the detection of abnormal masses including breast cancer. The Bexa™ device uses highly accurate pressure sensors to perform elastographic evaluation of breast tissue under light compression in conjunction with proprietary image processing algorithms to identify breast masses. The device is simple to use which allows consistent results to be produced by different examiners. The Bexa™ device, hereafter referred to as "Bexa" consists of a sensor module (similar in shape to a computer mouse) with a capacitive sensor array that is connected to a tablet computer to process and visualize the results. Bexa has 510(k) clearance (K181672) from the US Food and Drug Administration (FDA) as a pressure mapping system for documentation of CBE findings under its former commercial name, "SureTouch." Sure, Inc.'s proprietary sensor array technology and processing algorithms are ideally suited for application to detection of abnormal breast masses including cancer because the technology is low-cost, highly portable, free of radiation, and consistently adopted by women in all racial and ethnic communities. Logistically, it addresses several structural and cultural barriers that prevent mass adoption of screening for breast cancer.

The Clinical Use of the Bexa Breast Exam:

The majority of morbidity and mortality from breast cancer is caused by malignancies that present as solid tumors of the breast. The Bexa device produces a clear and accurate image of breast masses as small as 4mm (as measured by B-mode ultrasound) and misses between 6 and 11% of masses of all types. Mammography has a theoretical resolution of 5mm and misses 20% of breast cancers, and a higher proportion of all masses. Based on prior studies, Bexa is the best means of identifying solid masses in the breast including cancer.

In the U.S. population, Bexa will identify a mass in approximately 8%-11% of women, and these masses require additional evaluation. By comparison, mammography has a false-positive rate requiring 12%-14% of women to have unnecessary additional evaluation. The actual rate of referral for additional studies following screening mammography is often higher based upon claims review and not just false positive findings in the medical literature. As well, the literature demonstrates the known efficacy of mammography in women older than 50, with no effective solution available in the less than 50 population. Compared to mammography, the Bexa device used as an early detection technology improves mass detection accuracy while reducing the proportion of women referred for additional and unnecessary imaging studies and biopsies.

The results of the BBE are provided to women immediately whereas the results of screening mammogram examinations are require a subsequent, non-synchronous interpretation by a radiologist.

The most common next-step evaluation of a mass identified by Bexa is an ultrasound of the mass. Simple physiologic cysts and benign solid tumors can be easily identified by a focused or "spot," ultrasound of the detected mass. Based upon more than 500 masses identified by Bexa exams performed by ARDMS breast ultrasound technicians, up to half have been found to be easily identified as benign. This reduces the rate of women referred from a single visit consisting of a Bexa exam combined with "spot" ultrasound of discovered masses- to less than 4%, compared to greater than 12% referred for additional studies following a mammogram.

The Bexa Breast Exam process produces accuracy in mass identification that exceeds the limit of lesion size and depth detectable by conventional manual palpation techniques used during a Clinical Breast Exam and digital mammography. The Bexa Breast Exam similarly requires that a far smaller proportion of women examined require additional appointments and studies compared to women undergoing mammography.

Bexa has the potential to serve as an accurate, consistent, low-cost early detection modality that can be widely deployed in U.S. and global community settings, mobile units, as well as traditional and non-traditional primary care settings.

ELIGIBILITY:
Inclusion Criteria:

1. Women who present to receive a screening mammogram.
2. Women of all races, ethnicities, and socio-economic backgrounds.
3. Signed informed consent obtained prior to any study assessments and procedures.
4. Age 30-75 years of age and female.

Exclusion Criteria:

1. Women with findings that are < 0.5 cm or > 3.5 cm
2. Palpable lesion (to the participant)
3. Positive clinical findings that cause a visible and obvious deformity of the breast or alteration in the skin appearance of the breast.
4. Women with breast tenderness significant enough to prevent completion of any of the study examinations. (Both ultrasound and Bexa require a light degree of pressure on the breast; certain women, very few, have enough breast tenderness that they cannot tolerate the pressure of either Bexa or ultrasound. Mammograms exert substantially more pressure on the breast.)
5. Women with breast significant skin scarring enough to prevent effective BBE (e.g., keloid scarring of the breast, for example), because extensive, hard surface scarring introduces artifact in the Bexa exam. Participant exclusion will be determined by the Bexa examiner.
6. Greater than 3 positive findings in a given breast.
7. Women who are unable to comprehend or unwilling to sign an informed consent form.
8. Women ages < 30 and > 75 years of age.
9. Pregnant women.
10. Women who have had a mastectomy - unilateral or bilateral.
11. Women who have had a recent (past 30 days) biopsy performed.
12. Women who have had a prior history of breast cancer in either breast.
13. Women who have had radiation to the breast.
14. Women who have had any breast surgery within the last 12 months.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 500 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Bexa Sensitivity of Mass Detection | During procedure
  Bexa sensitivity of mass detection as compared to digital tomosynthesis mammography

SECONDARY OUTCOMES:
False Negative Comparison between Bexa and Mammography | During procedure
  Compare masses identified by one modality and missed by the other
Bexa Detected Breast Cancers | 8 weeks
  Determine how many masses detected by Bexa are biopsy-proven cancers

CONTACTS AND LOCATIONS:
Overall Officials: John Cole, DO, Principal Investigator — Hendrick Health
Locations (1):
- Hendrick Health - Vera West Women's Center, Abilene, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarvazyan A, Egorov V, Son JS, Kaufman CS. Cost-effective screening for breast cancer worldwide: current state and future directions. Breast Cancer (Auckl). 2008;1:91-9. doi: 10.4137/bcbcr.s774. Epub 2008 Jul 2. PMID 19578481
- [Background] Miglioretti DL, Lange J, van den Broek JJ, Lee CI, van Ravesteyn NT, Ritley D, Kerlikowske K, Fenton JJ, Melnikow J, de Koning HJ, Hubbard RA. Radiation-Induced Breast Cancer Incidence and Mortality From Digital Mammography Screening: A Modeling Study. Ann Intern Med. 2016 Feb 16;164(4):205-14. doi: 10.7326/M15-1241. Epub 2016 Jan 12. PMID 26756460
- See also: US Preventive Services — https://www.uspreventiveservicestaskforce.org/uspstf/recommendation/breast-cancer-screening
- See also: SEER — https://seer.cancer.gov/statfacts/html/breast.html